CLINICAL TRIAL: NCT03179787
Title: Post-Marketing Surveillance Study of Aripiprazole in Patients With Autism
Status: Completed | Type: Observational
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 031-101-00116
Record Dates: First submitted 2017-06-01; First posted 2017-06-07 (Actual); Results first posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Aripiprazole oral product — oral administration of aripiprazole

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of aripiprazole in patients with autism in the real world clinical setting in Japan.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as autism with irritability

Exclusion Criteria:

* patients who has ever been treated with aripiprazole

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: naive patients with aripiprasole
Sampling Method: Non-Probability Sample
Enrollment: 528 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pharmacovigilance, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Otsuka Pharmaceutical Co., Ltd., Tokyo, Japan

REFERENCES:
- [Derived] Sugimoto Y, Yamamura K, Takayama T, Fukuta Y, Aoki K, Mikami K, Tomoda A. Aripiprazole in the real-world treatment for irritability associated with autism spectrum disorder in children and adolescents in Japan: 52-week post-marketing surveillance. BMC Psychiatry. 2021 Apr 22;21(1):204. doi: 10.1186/s12888-021-03201-6. PMID 33888067

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This surveillance was conducted in 528 participants from 100 trial sites in Japan.
Pre-assignment Details: Patients newly treated with aripiprazole for irritability associated with autism spectrum disorder (ASD) in children and adolescents (≥6 years and <18 years) were included.
Groups:
- Safety Analysis Group: Five hundred and twenty-eight patients were enrolled at 100 sites across Japan, and 526 case reports were collected during the period of April 2017 to September 2019. The safety analysis population consisted of 510 patients. Among excluded patients, 15 patients were lost to follow-up, and one patient was not treated with aripiprazole.
Period: Overall Study
Arm/Group | Safety Analysis Group
Started | 528
Completed | 510
Not Completed | 18
Not completed — Lost to Follow-up | 15
Not completed — Case report failures | 2
Not completed — Treatment not administered | 1

BASELINE CHARACTERISTICS:
Arm/Group | Safety Analysis Group
Number analyzed (Participants) | 510
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 510
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.4 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134
  Male | 376
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 510
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Japan | 510

OUTCOME MEASURES:

1. Primary Outcome: Mean Changes of Aberrant Behavior Checklist-Japanese Version (ABC-J) Irritability Subscale Scores From Baseline.
Description: Using caregiver-rated ABC-J, the degree of aberrant behaviors was scored on four levels ranging from 0 'not at all a problem', 1 'slight problem', 2 'moderately serious problem' to 3 'the problem is severe in degree' in irritability subscale (including 15 items describing symptoms of irritability, such as temper tantrums, aggression, mood changes, and self-injury).
  The irritability subscale score ranging from 0 to 45 was derived from the sum of the 15 items and higher values represent a worse outcome.
Time Frame: Baseline, Week 4, 8, 16, 24, 52
Population: Twenty-one patients with the protocol deviations (including all effectiveness measures were not assessed after treatment: n = 11, all effectiveness measures were assessed over 7 days after last dose: n = 7, the daily dose was > 15 mg: n = 2, all effectiveness were assessed after day 393: n = 1) were excluded, and then efficacy sample consisted of all participants who have Baseline and at least one Post-Baseline effectiveness evaluation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Safety Analysis Group
Number analyzed (Participants) | 396
score on a scale
  Baseline | 19.8 (9.5)
  Week 4: number analyzed (Participants) | 288
  Week 4 | 14.7 (8.8)
  Week 8: number analyzed (Participants) | 316
  Week 8 | 12.9 (8.1)
  Week 16: number analyzed (Participants) | 302
  Week 16 | 12.7 (8.3)
  Week 24: number analyzed (Participants) | 291
  Week 24 | 13.4 (8.9)
  Week 52: number analyzed (Participants) | 205
  Week 52 | 13.1 (9.1)
  End-point (LOCF) | 13.0 (9.0)

ADVERSE EVENTS:
Time Frame: Adverse events were observed from first dose until follow-up for 52 weeks.
Description: The adverse events (if any occurred), onset date, seriousness, outcome, date of outcome, causality to aripiprazole, other possible causal factors, and treatment for adverse events during the observation period were recorded. Seriousness was determined by the physicians.
Arm/Group | Safety Analysis Group
All-Cause Mortality (participants affected / at risk) | 0/510
Serious Adverse Events (participants affected / at risk) | 3/510
Other Adverse Events (participants affected / at risk) | 82/510
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Analysis Group (N=510)
Epilepsy (Nervous system disorders) | 1 (1)
Partial seizures (Nervous system disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Impulsive behaviour (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Analysis Group (N=510)
Somnolence (Nervous system disorders) | 48 (48)
Weight increased (Investigations) | 18 (18)
Headache (Nervous system disorders) | 8 (8)
Nausea (Gastrointestinal disorders) | 7 (7)
Increased appetite (Metabolism and nutrition disorders) | 6 (6)
Obesity (Metabolism and nutrition disorders) | 5 (5)

LIMITATIONS AND CAVEATS:
It was an observational study in daily clinical practice without a comparison group. In addition, there were deficiencies in the assessments and variations in the reports and evaluation based on the reporting made by the physicians and caregivers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-12-06): https://cdn.clinicaltrials.gov/large-docs/87/NCT03179787/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-26): https://cdn.clinicaltrials.gov/large-docs/87/NCT03179787/SAP_001.pdf